CLINICAL TRIAL: NCT05376332
Title: Sonomyographic Upper Limb Prosthetics: A New Paradigm
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Collaborators: Infinite Biomedical Technologies (Industry); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1492070-2; 1U01EB027601 (NIH)
Record Dates: First submitted 2022-03-21; First posted 2022-05-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Amputation; Prosthesis User

STUDY DESIGN:
Intervention Model Description: Crossover model: Participants receive one of two alternative interventions during the initial phase of the study and receive the other intervention during the second phase of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sonomyographic control (Experimental): Sonomyographic control involves the use of ultrasound signals from muscle deformation to control a prosthetic hand.
  Interventions: Device: Sonomyographic Prosthesis
- Myoelectric control (Active Comparator): Myoelectric control involves the use of surface electromyography signals from muscle activation to control a prosthetic hand.
  Interventions: Device: Myoelectric direct control prosthesis; Device: Myoelectric pattern recognition prosthesis

INTERVENTIONS:
Device: Sonomyographic Prosthesis — The sonomyographic system will include a custom-fitted test socket incorporating ultrasound transducers and controlling a TASKA prosthetic hand. All socket fittings will be performed by a board-certified prosthetist as part of this study.
  Arms: Sonomyographic control
Device: Myoelectric direct control prosthesis — The direct control system will include a custom-fitted test socket incorporating dual-site electrodes and controlling a TASKA prosthetic hand. All socket fittings will be performed by a board-certified prosthetist as part of this study.
  Arms: Myoelectric control
Device: Myoelectric pattern recognition prosthesis — The pattern recognition system will include the subject's clinically-prescribed socket and commercially-available pattern recognition technology (IBT Sense). The pattern recognition system will not be fitted as part of this study, as subjects will already be trained users prior to enrolling in the study.
  Arms: Myoelectric control

SUMMARY:
The vast majority of all trauma-related amputations in the United States involve the upper limbs. Approximately half of those individuals who receive a upper extremity myoelectric prosthesis eventually abandon use of the system, primarily because of their limited functionality. Thus, there continues to be a need for a significant improvement in prosthetic control strategies.

The objective of this bioengineering research program is to develop and clinically evaluate a prototype prosthetic control system that uses imaging to sense residual muscle activity, rather than electromyography. This novel approach can better distinguish between different functional compartments in the forearm muscles, and provide robust control signals that are proportional to muscle activity. This improved sensing strategy has the potential to significantly improve functionality of upper extremity prostheses, and provide dexterous intuitive control that is a significant improvement over current state of the art noninvasive control methods. This interdisciplinary project brings together investigators at George Mason University, commercial partners at Infinite Biomedical Technologies as well as clinicians at MedStar National Rehabilitation Hospital.

The investigators will optimize and implement algorithms for real-time classification and control with multiple degrees of freedom (DOF) using a miniaturized ultrasound system incorporated into a prosthetic socket. The investigators will then compare control performance between and sonomyography and myoelectric control (both direct control and pattern recognition) using a virtual environment as well as for performance of tasks related to activities of daily living. The investigators have two specific aims.

Specific Aim 1: Compare between sonomyography and myoelectric direct control Specific Aim 2: Compare between sonomyography and pattern recognition with velocity control The successful completion of this project will lead to the first in human evaluation of an integrated prototype that uses low-power portable imaging sensors and real-time image analysis to sense residual muscle activity for prosthetic control. In the long term, the investigators anticipate that the improvements in functionality and intuitiveness of control will increase acceptance by amputees.

DETAILED DESCRIPTION:
Specific Aim 1: Compare between sonomyography and myoelectric direct control The investigators would like to test the null hypothesis that there is no difference in performance on virtual environment and clinical outcome measures between sonomyographic and direct myoelectric control with mode-switching.

Participants: The investigators will recruit a total of 10 unilateral trans-radial amputees based on the inclusion and exclusion criteria. These participants will be naïve to use of myoelectric prostheses. This study is focused on trans-radial amputees who represent the largest population of users.

Protocol:

After informed consent is obtained, the investigators will perform a baseline evaluation of the subject's functionality using the Orthotics and Prosthetics User Survey Upper Extremity Functional Status (OPUS-UEFS). Then subjects will be randomized to either the Experimental first group (sonomyography control) or Standard first group (direct control). Subjects will be tested using both control systems following a two-by-two AB/BA crossover design.

The sonomyographic system will include a custom-fitted test socket incorporating ultrasound transducers and controlling a TASKA prosthetic hand. The direct control system will include a custom-fitted test socket incorporating dual-site electrodes and controlling a TASKA prosthetic hand. All socket fittings will be performed by a board-certified prosthetist as part of this study.

After being fit with the sonomyography system, subjects in the Experimental first group will undergo 4 hours of standard occupational therapy training by a certified therapist. The training will be distributed over 2 days with 2 hours of training per day. At the end of each hour of training, subjects will perform a Fitts' Law task in a virtual environment. The task and the primary and secondary outcome measures are described below. After the training has been completed, subjects will evaluated using a series of primary and secondary clinical outcome measures, as described below. Finally, subjects will complete the Satisfaction with Prosthesis section of the Trinity Amputation and Prosthesis Scales - Revised (TAPES-R) to assess satisfaction with the sonomyography system. After a washout period of 4 weeks, subjects will cross-over to the Standard system. Subjects will be fitted with the direct control system and undergo the same training and testing procedure described above.

Subjects in the Standard first group will be trained and tested with the direct control system first, and then cross over to the sonomyography system.

Details of Fitts' Law task protocol:

Subjects will move their limb into one of 4 positions following a display indicated on a screen (Fig. 16 in Research Strategy). Achieving each target position requires a different amount of shoulder abduction. When participants have reached the required limb position, an annulus-shaped target will be displayed. Subjects will use their prosthesis to perform a Fitts' Law task that involves controlling the position and size of a ring-shaped cursor in order to match the target. The Fitts' Law task will have one, two, or three degrees of freedom, where each degree of freedom is mapped to a specific motor intent. For example, wrist flexion can control horizontal cursor movement, pronation/supination can control vertical cursor movement, and hand open/close can control the cursor's radius. Subjects will be allowed to activate the degrees of freedom sequentially or simultaneously.

The annulus width (W) and distance (D) from the initial cursor position will be varied to create six indices of difficulty according to ID = log2(1+ D/W). There will be three levels of target complexity based on the number of degrees of freedom that must be activated to achieve the task (i.e., one degree of freedom targets require activity in only one degree of freedom, etc.). Each possible combination of levels of difficulty (6) and target complexities (3) will be repeated 3 times per limb position.

Subjects will have 10 seconds to match the target and hold for two seconds, or the attempt will be considered failed. After 12 seconds, the display will indicate the next target.

Data Analysis:

Data will be evaluated to determine the distribution and the variability of performance within and between the different prosthesis systems. The investigators will test whether the sonomyography and direct control systems are equivalent using the primary outcome measures. Secondary outcome measures will also be explored in order to develop a more detailed understanding of differences in performance between the systems. If significant differences are found in baseline functional measures using OPUS-UEFS, the investigators will perform stratified analyses on our primary and secondary outcome measures.

Specific Aim 2. Compare between sonomyography and pattern recognition with velocity control Participants: The investigators will recruit a total of 6 unilateral trans-radial amputees based on the inclusion and exclusion criteria noted above. These participants will be experienced users of myoelectric pattern recognition control (IBT Sense). This study is focused on trans-radial amputees who represent the largest population of users.

Protocol:

After informed consent is obtained, the investigators will perform a baseline evaluation of the subject's functionality using the Orthotics and Prosthetics User Survey Upper Extremity Functional Status (OPUS-UEFS). Then subjects will be randomized to either the Experimental first group (sonomyography control) or Standard first group (pattern recognition control). Subjects will be tested using both control systems following a two-by-two AB/BA crossover design.

The sonomyographic system will include a custom-fitted test socket incorporating ultrasound transducers and controlling a TASKA prosthetic hand. All socket fittings will be performed by a board-certified prosthetist as part of this study. The pattern recognition system will include the subject's clinically-prescribed socket and commercially-available pattern recognition technology (IBT Sense). The pattern recognition system will not be fitted as part of this study, as subjects will already be trained users prior to enrolling in the study.

After being fit with the sonomyography system, subjects in the Experimental first group will undergo 4 hours of standard occupational therapy training by a certified therapist. The training will be distributed over 2 days with 2 hours of training per day. At the end of each hour of training, subjects will perform a Fitts' Law task in a virtual environment. The task and the primary and secondary outcome measures are described below. After the training has been completed, subjects will evaluated using a series of primary and secondary clinical outcome measures, as described below. Finally, subjects will complete the Satisfaction with Prosthesis section of the Trinity Amputation and Prosthesis Scales - Revised (TAPES-R) to assess satisfaction with the sonomyography system. After a washout period of 4 weeks, subjects will cross-over to the Standard system. Subjects will not undergo training, and will instead be immediately tested with the pattern recognition system using both the Fitts' Law task and clinical outcome measures.

Subjects in the Standard first group will be tested with the pattern recognition system first, and then cross over to the sonomyography system.

Data Analysis:

Data will be evaluated to determine the distribution and the variability of performance within and between the different prosthesis systems. The investigators will test whether the sonomyography and pattern recognition control systems systems are equivalent using the primary outcome measures. Secondary outcome measures will also be explored in order to develop a more detailed understanding of differences in performance between the systems. If significant differences are found in baseline functional measures using OPUS-UEFS, the investigators will perform stratified analyses on our primary and secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Transradial unilateral amputation
* Fluent in English
* For active comparator intervention 1 (myoelectric direct control prosthesis): Naïve to use of myoelectric prosthesis (i.e., uses body-powered prosthesis or has not used a myoelectric prosthesis for at least 3 years)
* For active comparator intervention 2 (myoelectric pattern recognition control prosthesis): Currently uses a commercially-available pattern recognition system (IBT Sense) with a terminal device having at least two degrees of freedom

Exclusion Criteria:

* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation
* Uncontrolled pain or phantom pain impacting full participation in the study as determined upon OT evaluation
* Serious uncontrolled medical problems as judged by the project therapist

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Fitt's Law Throughput | at one week
  The investigators will use throughput as the primary outcome measure for the Fitt's Law task. Throughput is defined as the ratio of index of difficulty to the movement time required for successful completion.
Southampton Hand Assessment Procedure (SHAP) | at two weeks
  The Southampton Hand Assessment Procedure (SHAP) will be the primary clinical outcome measure. The SHAP is a time-based test of a standardized protocol of 26 timed activities of daily living (ADL) tasks. The SHAP has a set of common objects representative of everyday items for the user to pick up. The results of the SHAP is a score which directly compares the abilities of the subject with those of intact able-bodied individuals as well as more refined scores for six prehensile patterns. A SHAP score of 100 is what an intact person is expected to achieve. Lower scores indicate worse function. This test has been validated for normative data.

SECONDARY OUTCOMES:
Fitt's Law Path Efficiency | at one week
  The investigators will use the path efficiency as a secondary outcome measure for the Fitt's Law task. Path efficiency is defined as the ratio of the shortest path to target and the actual path taken by the cursor for a successful completion. The path efficiency is a measure of the dexterity and intuitiveness of the control strategy.
Fitt's Law Completion Rate | at one week
  The investigators will use completion rate as a secondary outcome measure for the Fitt's Law task. Completion rate is defined as the percentage of targets that subjects can match and hold for 2 seconds within the allotted time. Target matching and holding is defined as staying within a 10% tolerance around the target.
Clothespin Relocation Test (CRT) | at two weeks
  The Clothespin Relocation Test (CRT) is a timed measure requiring users to grasp and move clothes pins, rotate the orientation of the clothes pins, and reposition them up and then back down a metal rod positioned at waist level.
Gaze and Movement Assessment (GaMA) | at two weeks
  The Gaze and Movement Assessment (GaMA) Protocol uses motion capture and eye tracking to quantify the movement and visual attention of participants as they perform object interaction tasks. The GaMA Protocol includes: (1) a procedure for the administration of two standardized functional tasks - the 'Pasta Box Task' and 'Cup Transfer Task'; (2) a methodology to obtain synchronized motion capture and eye tracking data during functional task execution; and (3) a data analysis software tool, which requires a standardized data set of synchronized movement and eye data coordinates as input, and outputs measures of hand movement, angular joint kinematics, and eye gaze. The protocol has been validated in the scientific literature and administered in prosthetic user populations. The GaMA metrics are quantitative measures of kinematics and eye movement. These metrics are not reported on a scale.
Satisfaction with Prosthesis section of the Trinity Amputation and Prosthesis Scales - Revised (TAPES-R) | Baseline
  The Trinity Amputation and Prosthesis Scales - Revised (TAPES-R) is a 33-item multidimensional questionnaire. The questionnaire has three sections: (1) psychosocial adjustment, which consists of three 5-item subscales: general adjustment. social adjustment, and adjustment to limitation; (2) activity restriction, which consists of ten items; and (3) satisfaction with the prosthesis section which consists of two subscales: aesthetic (3 items) and functional (5 items) satisfaction. The range of scores is 1-30. Higher scores are indicative of greater adjustment, lower activity restriction and more satisfaction with the prosthesis.
Orthotics and Prosthetics User Survey Upper Extremity Functional Status (OPUS-UEFS) | Baseline
  The Orthotics and Prosthetics User Survey Upper Extremity Functional Status (OPUS-UEFS) is a 23-item survey questionnaire designed to understand the subject's functional status at baseline. The range of scores is 0 - 92. A higher score indicates greater function.

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha Sikdar, PhD, Principal Investigator — George Mason University
Locations (1):
- Peterson Health Sciences Hall, Fairfax, Virginia, United States